CLINICAL TRIAL: NCT00189787
Title: Dose Response of Inhaled Tacrolimus in Patients With Moderate Persistent Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Astellas Pharma Europe B.V. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FG-506-17-07
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2008-04-17 (Estimated); Status verified 2008-04

CONDITIONS: Asthma, Bronchial; Bronchial Asthma
Keywords: Tacrolimus; Immunosuppressant; Anti-asthmatic drug; Administration, inhalation
MeSH Terms: conditions — Asthma; Respiratory Aspiration | interventions — Tacrolimus

INTERVENTIONS:
Drug: tacrolimus

SUMMARY:
This study will evaluate the efficacy and safety of tacrolimus in patients with asthma.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of asthma
* Patients treated with inhaled corticosteroid
* FEV1 (forced expiratory volume in 1 second)>60% to 80%

Exclusion Criteria:

* Respiratory infection within 2 weeks
* Asthma exacerbation within 90 days

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 370 (Actual)
Dates: Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: R.G.M.vom Amsterdam, MD, Study Director — Astellas Pharma Europe B.V.
Locations (37):
- Bulgaria (4):
  - Pleven
  - Rousse
  - Sofia
  - Varna
- Czechia (4):
  - Brno
  - Krhanice
  - Olomouc
  - Šumperk
- Germany (10):
  - Berlin
  - Bonn
  - Deggendorf
  - Düsseldorf
  - Hanover
  - München
  - Potsdam
  - Rüdersdorf
  - Solingen
  - Wiesbaden
- Hungary (5):
  - Budapest
  - Csorna
  - Füzesabony
  - Nyíregyháza
  - Szombathely
- Poland (6):
  - Bialystok
  - Krakow
  - Lodz
  - Lublin
  - Tarnów
  - Wroclaw
- Russia (5):
  - Moscow
  - Rostov-on-Don
  - Saint Petersburg
  - Smolensk
  - Yekaterinburg
- Ukraine (3):
  - Dnipro
  - Donetsk
  - Kiev